CLINICAL TRIAL: NCT02222090
Title: Therapy With New Oral Anticoagulants in Patients With Atrial Fibrillation and Renal Impairment
Brief Title: Therapy With New Oral Anticoagulants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-14-1181-IG-CTIL
Record Dates: First submitted 2014-08-04; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Atrial Fibrillation; Non-valvular Atrial Fibrillation
Keywords: patients with atrial fibrillation (AF) recommend the use of novel oral anticoagulants (NOACs) in patients with non-valvular AF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients who have been prescribed warfarin
- patients who have been prescribed apixaba

SUMMARY:
The aim of the present registry is to characterize and follow patients prospectively and retrospectively with renal impairment who have been prescribed apixaban for the prevention of stroke in atrial fibrillation, with a comparison to the characteristics and outcomes associated with warfarin therapy in this population.

DETAILED DESCRIPTION:
Current guidelines for the management of patients with atrial fibrillation (AF) recommend the use of novel oral anticoagulants (NOACs) in patients with non-valvular AF .Renal dysfunction has been shown to be an independent predictor of stroke or systemic emboli, but the risk of bleeding with conventional warfarin therapy is also significantly increased.Prevalence of renal dysfunction in patients with atrial fibrillation is high, with approximately 60% of patients having an estimated glomerular filtration rate (eGFR) of ≤ 60 ml/min/BSA [6].NOACs undergoing significant renal secretion such as dabigatran are not recommended for patients with severe renal impairment, and dose adjustment are indicated for patients with milder degrees of renal dysfunction.However, real-world information regarding the usage and outcomes associated with NOAC therapy in patients with renal dysfunction are limited. The investigators plan to prospectively and retrospectively collect data regarding the clinical settings, characteristics, and outcomes of patients with renal dysfunction who have been prescribed apixaban in Israel, using a multicenter secure web-based registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal dysfunction (eGFR <60 ml\min\BSA) who have an indication for treatment with an novel oral anticoagulant agent or VKA
* Patients prescribed apixaban or warfarin at the enrollment center (patients enrolled in a 2:1 ratio)

Exclusion Criteria:

* Valvular AF or presence prosthetic valve
* Dialysis patients
* Contraindications NOACs
* Hepatic dysfunction
* Cognitive impairment
* Clinical necessity to continue administration of potent inhibitors of both CYP3A4 and P-gp - including azole- antimycotics (e.g. ketoconazole, itraconazole) and HIV protease inhibitors (e.g. ritonavir)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients prospectively and retropectively with renal impairment who have been prescribed apixaban for the prevention of stroke in atrial fibrillation, with a comparison to the characteristics and outcomes associated with warfarin therapy in this population
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes | within 12 month from enrollment
  To evaluate the clinical characteristics, treatment indications, and risks of stroke and bleeding in non-valvular atrial fibrillation patients prescribed apixaban or warfarin.

SECONDARY OUTCOMES:
one-year outcomes | within 12 month from enrollment
  Establish the one-year outcomes of this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, Prof, Study Director — Sheba Medical Center; Alon Barsheshet, MD, Principal Investigator — beilinson Medical Center; Avishay Elias, MD, Principal Investigator — beilinson Medical Center; Shmuel Fuchs, Prof, Principal Investigator — beilinson Medical center; KIRILL BUTURLIN, MD, Principal Investigator — Meir Medical Center; Moshe Swissa, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel